CLINICAL TRIAL: NCT02172547
Title: Effect of Spiriva® 18 Microgram on Health-related Quality of Life in COPD Patients Who Stopped Smoking During Treatment.
Brief Title: Effect of Spiriva® on Health-related Quality of Life in Chronic Obstructive Pulmonary Disease (COPD) Patients Who Stopped Smoking During Treatment.
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.364
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- COPD patients who stopped smoking during treatment
  Interventions: Drug: Spiriva

INTERVENTIONS:
Drug: Spiriva

SUMMARY:
Post marketing Surveillance to gain insights into the effects of therapy with Spiriva® (tiotropium bromide) on health-related quality of life in COPD patients who stopped smoking during treatment and to obtain safety data regarding adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD
* Smoker at start

Exclusion Criteria:

* Patients presenting with any general and specific contraindications listed in the Patient Information Leaflet ('Gebrauchsinformation') and the Basic Product Information('Fachinformation')

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Practioner
Sampling Method: Non-Probability Sample
Enrollment: 10821 (Actual)
Dates: Start 2006-04; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Changes in health related quality of life | 6 weeks

SECONDARY OUTCOMES:
Occurrence of Adverse events | 6 weeks